CLINICAL TRIAL: NCT02722889
Title: Ascending Aortic Length in Relation to Age and the Occurrence of Type A Aortic Dissection
Brief Title: Aortic Elongation and Dissection
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-4-027
Record Dates: First submitted 2016-03-07; First posted 2016-03-30 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2016-03

CONDITIONS: Thoracic Aorta
Keywords: Ascending aorta; Elongation of the aorta; Type A dissection; Aortic rupture; Aortic length
MeSH Terms: conditions — Aortic Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy controls: Healthy control patients
- Type A dissection: Patients with proven type A dissection,

SUMMARY:
Aim of this study is to measure length of the ascending aorta in adults and to investigate the clinical implication of 'elongation' of the aorta.

DETAILED DESCRIPTION:
Regarding to aortic geometry, attention is often drawn to aortic diameters since an increase in these diameters (e.g. aneurysm) can lead to life-threatening complications such as dissection and/or rupture. In daily practice however (e.g. imaging reports), the investigators often encounter patients with elongation of the ascending aorta. Little is known about the length of the proximal aorta. Furthermore, the clinical implications of an elongated aorta are unknown.

ELIGIBILITY:
Inclusion Criteria:

* Underwent recent (<6 years) contrast-enhanced CT scan which allows for segmentation and assessment of aortic geometry.

Exclusion Criteria:

* Age <18 years old.
* Prior thoracic, cardiac or aortic surgery.
* Genetic disease with cardiac and/or aortic involvement (e.g. Marfan's disease).
* Infectious disease of the aorta.
* Malignant disease with involvement of heart and/or aorta.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Reference group to assess 'normal' aortic length.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Length of the ascending aorta | Up to 72 months
  Ascending aortic length as measured on computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wildberger, MD, PhD, Principal Investigator — Head of department of Radiology
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No